CLINICAL TRIAL: NCT06561945
Title: Accuracy of Dental Movements Using Clear Aligners Treatment: a Single-center Prospective Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Giorgio Gastaldi, Associate Professor, IRCCS Ospedale San Raffaele
Other Study IDs: CA-001
Record Dates: First submitted 2024-07-14; First posted 2024-08-20 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Malocclusion
Keywords: clear aligner; malocclusion; direct print aligner
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- orthodontic patients: Patients who need orthodontic treatment.

SUMMARY:
The aim of the present prospective observational study is to evaluate the accuracy of dental movements in the three planes of space, assessing the correspondence between the virtual planned movements and the clinical outcomes achieved using thermoformed or 3D printed orthodontic aligners. The study will include patients who are candidates for aligner orthodontics treatment. After having acquired the standard initial diagnostic data (clinical examination, intra- and extra-oral photographs, intra- and extra-oral scans, orthopantomography and lateral-lateral teleradiography of the skull), the digital impressions of the arches will be used to plan the dental movements necessary for correction of malocclusion.

The aligners will then be designed using orthodontic CAD software and realized using a thermoformed and direct 3D printing process.

All patients will be treated following current recommendations relating to the orthodontic treatments in question. After delivery of the aligners, during each check-up, intra-oral and extra-oral scans will be acquired to evaluate the actual position of the teeth and, using special software will be compare the virtually designed position with tooth with the clinical outcomes. Any discrepancies will be recorded and statistically analyzed.There are no additional invasive procedures. Intra- and extra-oral scans will be acquired regularly to monitor the extent of tooth movement over time.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years
2. Good general health
3. Presence of a dental/skeletal malocclusion
4. Permanent dentition with second molars completely erupted in the arch
5. Correct tooth shape, with sufficient height of the clinical crowns
6. Good compliance during treatment

Exclusion Criteria:

1. Systemic diseases or pharmacological therapy with drugs that can affect orthodontic movement
2. Orofacial malformations or syndromes
3. Periodontal disease
4. Smoke
5. Pregnancy
6. Signs and/or symptoms of temporomandibular disorders
7. Absence of teeth (except for third molars)
8. Dental Implants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from patients aged 18 years and older who require orthodontic treatment with clear aligners. One hundred patients will be enrolled, without distinction based on gender.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate accuracy aligners of on transversal dental linear movements | 18 months
  Correspondence between virtual planned linear movements (in millimetres) and clinical outcomes achieved using aligners evaluated on the transversal plane. Post-treatment digital models and final virtual treatment plan models will be exported as STL files and subsequently imported into Geomagic Qualify ®software, to compare final teeth positions
Evaluate accuracy aligners of on vertical dental linear movements | 18 months
  Correspondence between virtual planned linear movements (in millimetres) and clinical outcomes achieved using aligners evaluated on the vertical plane. Post-treatment digital models and final virtual treatment plan models will be exported as STL files and subsequently imported into Geomagic Qualify ®software, to compare final teeth positions
Evaluate accuracy aligners of on sagittal dental linear movements | 18 months
  Correspondence between virtual planned linear movements (in millimetres) and clinical outcomes achieved using aligners evaluated on the sagittal plane. Post-treatment digital models and final virtual treatment plan models will be exported as STL files and subsequently imported into Geomagic Qualify ®software, to compare final teeth positions

SECONDARY OUTCOMES:
Evaluate accuracy of 3d printed aligners on transversal dental angular movements | 18 months
  Correspondence between virtual planned angular movements (in degrees) and clinical outcomes achieved using aligners evaluated on the transversal plane. Post-treatment digital models and final virtual treatment plan models will be exported as STL files and subsequently imported into Geomagic Qualify ®software, to compare final teeth positions
Evaluate accuracy of 3d printed aligners on sagittal dental angular movements | 18 months
  Correspondence between virtual planned angular movements (in degrees) and clinical outcomes achieved using aligners evaluated on the sagittal plane. Post-treatment digital models and final virtual treatment plan models will be exported as STL files and subsequently imported into Geomagic Qualify ®software, to compare final teeth positions
Evaluate accuracy of 3d printed aligners on vertical dental angular movements | 18 months
  Correspondence between virtual planned angular movements (in degrees) and clinical outcomes achieved using aligners evaluated on the vertical plane. Post-treatment digital models and final virtual treatment plan models will be exported as STL files and subsequently imported into Geomagic Qualify ®software, to compare final teeth positions

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Gastaldi, MD, DDS, Principal Investigator — Vita-Salute San Raffaele University Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ferlias N, Dalstra M, Cornelis MA, Cattaneo PM. In Vitro Comparison of Different Invisalign(R) and 3Shape(R) Attachment Shapes to Control Premolar Rotation. Front Bioeng Biotechnol. 2022 Mar 16;10:840622. doi: 10.3389/fbioe.2022.840622. eCollection 2022. PMID 35372304
- [Result] Grunheid T, Loh C, Larson BE. How accurate is Invisalign in nonextraction cases? Are predicted tooth positions achieved? Angle Orthod. 2017 Nov;87(6):809-815. doi: 10.2319/022717-147.1. Epub 2017 Jul 7. PMID 28686090
- [Result] Houle JP, Piedade L, Todescan R Jr, Pinheiro FH. The predictability of transverse changes with Invisalign. Angle Orthod. 2017 Jan;87(1):19-24. doi: 10.2319/122115-875.1. Epub 2016 Jun 15. PMID 27304231
- [Result] Kravitz ND, Kusnoto B, BeGole E, Obrez A, Agran B. How well does Invisalign work? A prospective clinical study evaluating the efficacy of tooth movement with Invisalign. Am J Orthod Dentofacial Orthop. 2009 Jan;135(1):27-35. doi: 10.1016/j.ajodo.2007.05.018. PMID 19121497
- [Result] Papadimitriou A, Mousoulea S, Gkantidis N, Kloukos D. Clinical effectiveness of Invisalign(R) orthodontic treatment: a systematic review. Prog Orthod. 2018 Sep 28;19(1):37. doi: 10.1186/s40510-018-0235-z. PMID 30264270